CLINICAL TRIAL: NCT01819064
Title: Do Small Doses of Atropine Cause Bradycardia in Young Children
Brief Title: Heart Rate Response to Atropine Doses Less Than 0.1mg IV to Anesthetized Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesiology, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Atropine in infants
Record Dates: First submitted 2013-02-04; First posted 2013-03-27 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Bradycardia; Arrhythmias
Keywords: Atropine; bradycardia; tachycardia
MeSH Terms: conditions — Bradycardia; Arrhythmias, Cardiac; Tachycardia | interventions — Atropine

STUDY DESIGN:
Intervention Model Description: This is a single arm study where a dose of atropine was administered and the ECG recorded.
Masking Description: Observer of ECG rhythm strips was unaware of the study hypothesis, the study drug administered, the dose given and the arrhythmias sought. Your statement that masking a single outcome implies a multi-arm study precludes a panoramic perspective of clinical research study designs and scenarios in which assessors may be effectively blinded.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Infants and children less than 15Kg. (Experimental): This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure and weigh less than 15Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
  Interventions: Drug: Atropine

INTERVENTIONS:
Drug: Atropine — intravenous atropine affect on heart rate
  Other Names: atropine sulfate; atropine injection

SUMMARY:
An infants heart rate is very important because it ensures that blood is pumped to all organs in the body. Heart rate may decrease during anesthesia and surgery, and this is why the anesthesiologist will often give a medication to prevent this from happening. The most common drug for this purpose is called atropine. The dose of most drugs given to babies is based upon the baby's weight, but some believe that the dose of atropine should not be less than 0.1mg. However there is no evidence to support this minimum dose. A larger dose of atropine may cause a very fast heart rate instead. Anesthesiologists routinely dose the atropine based upon the baby's weight without regard for a minimum dose.

The purpose of the present study is to measure the heart rate after doses of atropine in neonates and infants who receive less than 0.1 mg.

DETAILED DESCRIPTION:
60 infants, ASA physical status I and II, undergoing elective surgical procedures will be enrolled after signed informed parental consent.

All children will be fasted according to institutional guidelines and unpremedicated. After arriving in the operating room, EKG, pulse oximeter and blood pressure monitors will be applied (Datex-Ohmeda Aisys).

Anesthesia will be induced with 66% N2O in O2 and 8% sevoflurane. Respiration will be supported by a properly sized face mask through which he/she is allowed to breath spontaneously. Respiration will continue spontaneously through a facemask at 2 MAC sevoflurane in 66% N2O.

All children will be positioned supine, warmed with a forced air warmer and given 20 ml/kg IV balanced salt solution over 30 minutes after the IV has been established. The end-tidal pCO2 will maintained 35-45 mmHg and oxygen saturation >96%.

After a 22 or 24G IV cannula is inserted, 0.005 mg/kg atropine will be administered intravenously over 5 seconds through a fast-flowing IV and followed by 5 ml of normal saline to flush it in through the IV deadspace. The study (ECG recording) period will extend from 30 seconds before atropine administration to 5 minutes after injection. During this time the heart rate and rhythm (through lead II) will be monitored and recorded continuously using an analogue interface system. EKG will be recorded on paper continuously for the 330 seconds of the study.

The recording will be analyzed for the heart rate (based on the R-R interval) and arrhythmias by a physician blinded to the study. Blinding means that the individual is unaware of the hypothesis of the study and what medication was administered to account for any changes in heart rate. Bradycardia is defined as a 20% reduction from baseline heart rate while tachycardia is a heart rate > 160 beats/minute(6). Any heart rate < 100/minute will be considered a bradycardia in this age group. Arrhythmia is any disorder of rhythm or rate observed. These will be summarized for each child.

All heart rate responses will be recorded and reviewed. The time to record the heart rate after atropine, which will occur before surgery, will add less than 5 additional minutes to the anesthetic since it will overlap the time taken for other surgical preparatory events.

The blood pressure will be monitored non-invasively immediately before receiving atropine and at one and five minutes after it is given.

The primary outcome is the incidence of bradycardia during the first 5 minutes after atropine will be determined by reviewing the electrocardiogram. All continuous data will be reported as means +/- standard deviation.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 0-2 years old
2. Weight : less than the 95th percentile for age and height ( no more than 15kg )
3. ASA classification : I-II
4. Meets the hospital and department of anesthesiology guidelines with respect to peri-operative care

Exclusion Criteria:

1. History of heart disease
2. Any condition predisposing to arrhythmia
3. Any medication known to influence the heart rate
4. Child taking anti-cholinergic medication routinely
5. The use of succinylcholine anticipated (will cause bradycardia)
6. Rapid sequence intubation is required (due to aspiration risk)
7. Known difficult airway (may be difficult to bag mask ventilate)

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD FRCPC, Principal Investigator — SUNY at Buffalo, Women and Children's Hospital of Buffalo
Locations (1):
- Women and Children's Hospital of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eisa L, Passi Y, Lerman J, Raczka M, Heard C. Do small doses of atropine (<0.1 mg) cause bradycardia in young children? Arch Dis Child. 2015 Jul;100(7):684-8. doi: 10.1136/archdischild-2014-307868. Epub 2015 Mar 11. PMID 25762533

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Weighing Less Than 15Kg: This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure and weigh less than 15Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
  Atropine: IV dose at 5 mcg/kg
Period: Overall Study
Arm/Group | Children Weighing Less Than 15Kg
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This was not a randomized or controlled variable
Groups:
- Children Less Than 15Kg.: This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure, and weighed less than 15Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
Arm/Group | Children Less Than 15Kg.
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 60
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: months] — age will be measured in months
  months | 6.5 [4 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 60
weight [Median (Inter-Quartile Range); unit: kilograms] | 8.1 [7.5 to 8.8]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Bradycardia
Description: incidence of bradycardia or other arrhythmias
Time Frame: five minutes
Population: There was no restriction on enrollment so long as the child was <15 kg.
Measure: Number; unit: participants
Groups:
- Children Less Than 5Kg.: This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure, and weighed less than 5Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
- Children Weighing 5Kg to 15Kg: This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure, and weighed between 5Kg and 15Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
Arm/Group | Children Less Than 5Kg. | Children Weighing 5Kg to 15Kg
Number analyzed (Participants) | 9 | 51
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: until the child is discharged from hospital on the day anesthesia was provided
Groups:
- Children Less Than 15Kg.: This group consists of children who are ASA physical status I and II, less than 2 years of age and scheduled for elective surgical procedure and weigh less than 5Kg will receive atropine 5 mcg/kg IV during sevoflurane anesthesia.
  Atropine: IV dose at 5 mcg/kg
Arm/Group | Children Less Than 15Kg.
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children Less Than 15Kg. (N=60)
asystole (Cardiac disorders) | 0 (0) — very slow heart rates, abnormal heart rhythms
asystole (Cardiac disorders) | 0 (0) — zero heart rate after low dose atropine in the five minutes after administration of atropine.
Bradycardia (Cardiac disorders) | 0 (0) — Slow or absent heart rate
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Children Less Than 15Kg. (N=60)
arrhythmias (Cardiac disorders) | 0 — atrial extrasystoles, bradycardia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No